CLINICAL TRIAL: NCT06338618
Title: Manual Therapy Effects in Patients With Metabolic-associated Fatty Liver Disease
Brief Title: Manual Therapy in Metabolic Liver Disease
Acronym: OSTEO-EHMet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Angel Oliva Pascual-Vaca, Head of Physiotherapy Department, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1532-N-23
Record Dates: First submitted 2024-03-15; First posted 2024-03-29 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: NAFLD, Non-alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- liver treatment protocol (Experimental): The liver treatment protocol consists of performing twelve visceral manual techniques in an approximate time of 30 minutes twice a week for 4 weeks.
  Interventions: Procedure: liver treatment protocol
- placebo comparator (No Intervention): This group will not receive any type of treatment

INTERVENTIONS:
Procedure: liver treatment protocol — The liver treatment protocol consists of performing twelve visceral manual techniques in an approximate time of 30 minutes twice a week for 4 weeks
  Arms: liver treatment protocol

SUMMARY:
Hepatic steatosis is a disease that is becoming more common in our society; approximately 40% of the population suffers from non-alcoholic fatty liver. The beneficial effect of manual therapy for the treatment of viscera dysfunctions such as the stomach or colon is known. The objective of this study is to demonstrate the anti-inflammatory effects of visceral manual therapy in patients with metabolic liver disease associated with non-alcoholic fatty liver.

DETAILED DESCRIPTION:
Chronic liver diseases such as metabolic disease associated with nonalcoholic fatty liver lead to a stiff liver due to activation of hepatic stellate cells or portal fibroblasts into matrix-producing myofibroblasts. Congested livers tend to fibrosis, while the physiological forces that the liver receives during physical activity and deep breathing could have a beneficial effect on it, favoring physiological remodeling.

The importance of the mobility of the viscera for their proper functioning is known. Likewise, the beneficial effect of physical activity on the liver is known. This physical activity includes a component of applying pressure on the liver. These pressures are also exerted during the techniques described for manual liver treatment. Although there is some evidence about the effectiveness of these manual techniques for the treatment of pain situations, the effect they could have on liver parameters is unknown.

For all these reasons, we aim to know the effect of manual liver techniques on biochemical and mechanical sensitivity parameters in subjects with Metabolic Disease Associated with Non-Alcoholic Fatty Liver (NAFLD).

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age with MetHD defined by an ultrasound compatible with hepatic steatosis and an HSI > 36

Exclusion Criteria:

* Fibrosis defined by FIB-4 > 2.67
* Hepatic cirrhosis
* Geographic dispersion to avoid losses
* Contraindication to manual therapy
* Diabetes mellitus tiype 1
* Severe hypertriglyceridemia with TG > 500 mg/dl at the time of recruitment
* Life expectancy less than one year
* Advanced chronic kidney disease (stage G4)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2024-04-03 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2024-09-20 (Actual)

PRIMARY OUTCOMES:
Hepatic steatosis index | Pre-intervention. Post-intervention 4 weeks
  Decrease in the hepatic steatosis index

SECONDARY OUTCOMES:
FIB-4 index | Pre-intervention. Post-intervention 4 weeks
  Decrease in the FIB-4 index
NAFLD-fibrosis index | Pre-intervention. Post-intervention 4 weeks
  Decrease in the NAFLD-fibrosis index
HOMA index | Pre-intervention. Post-intervention 4 weeks
  Decrease in the HMA index
TyG index | Pre-intervention. Post-intervention. 4 weeks
  Decrease in the TyG index
Change from baseline in algometry | Pre-intervention Post-intervention 4 weeks
  Pressure pain threshold in face and neck tissues. PPT levels defined as the minimum necessary
Visual analogue Scale | Pre-intervention. Post-intervention 4 weeks
  Self-perceived pain intensity

CONTACTS AND LOCATIONS:
Overall Officials: Angel Oliva Pascual-Vaca, Dr, Study Director — University of Seville
Locations (1):
- Universitary Hospital Juan Ramón Jiménez, Huelva, Spain

IPD SHARING:
Plan to Share IPD: No